CLINICAL TRIAL: NCT02270749
Title: Vitamin Deficiencies and Suppletion in Morbid Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VITAALII
Record Dates: First submitted 2014-10-09; First posted 2014-10-21 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Vitamin B12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Hydroxocobalamin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydroxocobalamin injection (Active Comparator): 25 patients receive the standard treatment of a vitamin B12 deficiency: hydroxocobalamin injection
  Interventions: Drug: Hydroxocobalamin
- FitForMe vitamin B12 tablets (Active Comparator): 25 patients receive a daily dose vitamine B12 tablets
  Interventions: Drug: FitForMe vitamin B12

INTERVENTIONS:
Drug: Hydroxocobalamin — patients are treated for 6 months with hydroxocobalamin. Patients will be treated with once a dose of 2000ug, after that treatment will be continued with a dose of 1000ug per 2 months. At timepoint 0, 2, 4 and 6 months after treatment vitamin B12 will be measured. At timepoint 0 and 6 also homocystein and methylmalonic acid will be measured.
  Arms: hydroxocobalamin injection
Drug: FitForMe vitamin B12 — patients are treated for 6 months with a daily dose of 1000ug vitamin B12 tablets. At timepoint 0, 2, 4 and 6 months after treatment vitamin B12 will be measured. At timepoint 0 and 6 also homocystein and methylmalonic acid will be measured.
  Arms: FitForMe vitamin B12 tablets

SUMMARY:
The purpose of this study is to evaluate the most effective treatment for patients who underwent a Roux-en-Y gastric bypass and developed postoperatively a vitamin B12 deficiency.

DETAILED DESCRIPTION:
Vitamin B12 deficiency accounts up to 23-64% bariatric surgery. The investigators purpose is to evaluate the most effective treatment for vitamin B12 deficiency in patients who underwent a Roux-en-Y gastric bypass.

Daily oral use of vitamin B12 tablets are may be as effective as vitamin B12 injections.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin B12 deficiency: <200 pmol/l
* Vitamin B12 deficiency 6-12 months after surgery
* All patients underwent a Roux-en-Y gastric bypass

Exclusion Criteria:

1. Creatin >150micromol/L
2. Liver enzymes >2 times upper limit
3. Other bariatric operations
4. Intercurrent diseases
5. Gastro-intestinal diseases
6. Psychiatric disease
7. Medicines which influences bone density
8. Pregnancy

Ages: 18 Months to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
reduction in patients with vitamin B12 deficiency | 6 months after initiating therapy
  Before starting treatment vitamin B12, homocystein and methylmalonic acid will be measured. Two and 4 months after starting treatment vitamine B12 levels will be measured. At 6 months after initiating therapy again vitamin B12, homocystein and methylmalonic acid will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate hospital, Arnhem, Netherlands

REFERENCES:
- [Derived] Schijns W, Homan J, van der Meer L, Janssen IM, van Laarhoven CJ, Berends FJ, Aarts EO. Efficacy of oral compared with intramuscular vitamin B-12 supplementation after Roux-en-Y gastric bypass: a randomized controlled trial. Am J Clin Nutr. 2018 Jul 1;108(1):6-12. doi: 10.1093/ajcn/nqy072. PMID 29931179